CLINICAL TRIAL: NCT03391505
Title: Acute Effects of Physical Activity On Memory, Cognitive Performance and Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Krustrup, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 59349 to H-16026885
Record Dates: First submitted 2017-12-21; First posted 2018-01-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Mental Health Wellness 1
Keywords: Cognition; Physical activity; Memory; Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group 1 (Experimental): The small-sided soccer game consists of a single bout (two times ten minutes) of small-sided soccer game (3v3) interspersed with a five minutes break.
  Interventions: Behavioral: Small-sided soccer game
- Treatment Group 2 (Experimental): The walking soccer game consists of a single bout (two times ten minutes) of small-sided walking soccer game (3v3) interspersed with a five minutes break.
  Interventions: Behavioral: Walking soccer game
- Control Group (Placebo Comparator): The rest group watching soccer consists of watching a soccer game on a laptop (two times ten minutes) interspersed with a five minutes break.
  Interventions: Behavioral: Rest group watching soccer

INTERVENTIONS:
Behavioral: Small-sided soccer game — The small-sided soccer game consists of a single bout (two times ten minutes) of small-sided soccer game (3v3) interspersed with a five minutes break.
  Other Names: SSG
  Arms: Treatment Group 1
Behavioral: Walking soccer game — The walking soccer game consists of a single bout (two times ten minutes) of small-sided walking soccer game (3v3) interspersed with a five minutes break.
  Other Names: WSG
  Arms: Treatment Group 2
Behavioral: Rest group watching soccer — The rest group watching soccer consists of watching a soccer game on a laptop (two times ten minutes) interspersed with a five minutes break.
  Other Names: RES
  Arms: Control Group

SUMMARY:
The overall aim of the study is to investigate the effects of an acute bout of physical activity on cognitive performance and long-term memory in elementary school children. Elaborating, the study seeks to investigate the effect of the intensity of the physical activity on cognitive performance and long-term memory in preadolescent children.

DETAILED DESCRIPTION:
Based on a power analysis a total population of 100 children (four school classes) will be invited to participate in a 10-day protocol. The children will be randomly allocated, within their cluster (classes) and stratified for gender and soccer level, to one of 3 intervention groups. The groups consist of: A small-sides soccer game group (SSG), a walking soccer group (WSG) and a rest group watching soccer on TV (RES). At day 1 the children will complete a screening of their physical characteristics (height, weight, fat percentages, lean muscle mass and fitness status). On day 2 the children will complete a screening and a familiarization to the cognitive tasks used (cognitive performance and long-term memory) and the brain activity measuring devices (transportable EEG systems). On day 3 the children will complete the interventions, which first consist a long-term memory task, where the children will be asked to remember forty different pictures. Immediately after exposure to the forty pictures, the children will participate in 2 x 10 minutes of their respective interventions with 5 minutes break in between. During the break, the children will complete a short questionnaire to address their flow. Furthermore, during the intervention they will be equipped with heart rate monitors to quantify the physical demands of the intervention. Immediately after completing the 2 x 10 minutes interventions the children will be equipped with a transportable EEG system, and undergo a cognitive test (the Flanker task) to address their cognitive performance. The EEG recordings are used to measure the P3 amplitude and latency, biomarkers for cognitive performance. While equipping the children with the EEG system, the children will complete questionnaires about their participation. At day 10 the children will try to remember as many pictures of the forty pictures as possible to address the effect of the interventions on their long-term memory.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from the childrens´ legal guardians.
* Physical, linguistic and mental competencies to complete the intervention and testing.

Exclusion Criteria:

* Use of prescription-only drugs that kan affect learning ability.
* Smoking.
* Neurological diseases inclusive damages to the spinal cord.
* Children who is not evaluated to being cable of completing the protocol among these psychological diseases or psychological unstable children.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Event-related brain potentials (P300) | 1 day
  Electroencephalographic measures (mV) of the neuroelectric system that occur in response to, or in or in preparation for, a discrete event.
Cognitive Response Speed Performance | 1 day
  Measures of response speed (ms) during the computer-based Flanker task
Cognitive Response Accuracy Performance | 1 day
  Measures of response accuracy (%) during the computer-based Flanker task
Long-term Memory Accuracy Performance | 7 days
  Measures of response accuracy (%) during a tablet-based visual memory task

SECONDARY OUTCOMES:
Height | 1 day
  Measures of height (cm) with a Tanita Leicester portable altimeter
Weight | 1 day
  Measures weight (kg) with an InBody 230 multifrequency body composition analyser
Fat Percentage | 1 day
  Measures fat percentage (%) with an InBody 230 multifrequency body composition
Lean Body Mass | 1 day
  Measures of lean body mass (kg) with an InBody 230 multifrequency body composition
Fitness Status | 1 day
  Measures of distance covered during an maximal exercise test
Maximal Heart Rate | 1 day
  Measures of maximal heart rate with heart rate monitors during an maximal exercise test
Flow | 1 day
  Measures of flow with a danish translation og the flow questionnaire (Rheinberg et al., 2003) during the intervention
Motivation | 1 day
  Measures of motivation with the Intrinsic Motivation Inventory (IMI) questionnaire (McAuley et al., 1987) after the intervention
Enjoyment | 1 day
  Measures of self-perceived enjoyment with the Physical Activity Enjoyment Scale (PACES) (Kendzierski et al., 1991) questionnaire after the intervention
Intervention intensity | 1 day
  Measures of heart rate with heart rate monitors during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter Krustrup, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No